CLINICAL TRIAL: NCT01341067
Title: Continuous Glucose Monitoring in Subjects With Type 2 Diabetes
Brief Title: Continuous Glucose Monitoring (CGM) in Subjects With Type 2 Diabetes
Acronym: DexlonT2
Status: Completed | Type: Observational
Sponsor: Rocky Mountain Diabetes and Osteoporosis Center (Industry)
Responsible Party: Principal Investigator, David Liljenquist, M.D., Primary Investigator, Rocky Mountain Diabetes and Osteoporosis Center
Other Study IDs: RMDC-001
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Basal insulin, approved oral medications

SUMMARY:
The purpose of this study is to examine the effect CGM (continuous glucose monitoring) has on subjects with type 2 diabetes. It is anticipated that patients using the device will obtain tighter control of their blood sugars resulting in measureable health benefits and improved confidence in their ability to manage their diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with type 2 diabetes mellitus
* Have an HgbA1c value ≥ 7% and ≤17%.
* Are on basal insulin, with or without oral agents
* Are not on basal bolus insulin therapy.
* Have had no severe hypoglycemic episodes in the 6 months prior to enrollment in the study. Severe hypoglycemia will be defined as any hypoglycemia that is both neurologically impairing and absolutely requires assistance from a third party in the form of carbohydrates, glucagon shots, or attention from a paramedic or other healthcare professional.
* Have no known allergy to medical tape or sensors.
* Are capable of and willing to test their blood glucose (BG) on an average of 4 times per day.
* Are willing to not use Acetaminophen while enrolled in the study.
* Are willing not to undergo a MRI procedure while wearing the CGM sensor.
* Are willing and capable of performing self insertions of the device sensor.
* Women of child bearing potential must be willing to use an approved form of birth control while enrolled in the study.
* Women of child bearing potential must be willing to perform pregnancy tests monthly while enrolled in the study.
* Can understand and speak English fluently.

Exclusion Criteria

* Have been on pump therapy in the 6 months prior to enrollment in the study.
* Are receiving basal- bolus insulin therapy
* Are taking any medication that is not approved to be taken with insulin.
* Are pregnant or have intentions of becoming pregnant during the duration of the study.
* Have any skin condition that would inhibit the proper wearing of the CGM sensor including severe psoriasis, burns, eczema, scarring, excessive tattoos, etc.
* Have a hematocrit ≤30% or ≥55%
* Are currently enrolled in another clinical study (subjects must have ended participation in other studies at least 30 days prior to enrolling in this study.
* Are employed by any company that manufactures or is developing a CGM device.
* Are deemed incapable of participating in the study by the Primary Investigator for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of all adult ages (18 and older) with type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Liljenquist, MD, Principal Investigator — Rocky Mountain Diabetes and Osteoporosis Center
Locations (1):
- Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Basal Insulin, Approved Oral Medications: Basal insulin, with or without approved oral agents
Period: Overall Study
Arm/Group | Basal Insulin, Approved Oral Medications
Started | 30
Completed | 26
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Basal Insulin, Approved Oral Medications
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in HgbA1c
Time Frame: Measured at 6 months
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Basal Insulin, Approved Oral Medications
Number analyzed (Participants) | 26
percentage of glycosylated hemoglobin | -1.9 (1.1) [-3.0 to -.8]

2. Secondary Outcome: Percentage of Time Spent at Glycemic Levels <65 mg/dl
Time Frame: Measured at baseline and at 6 months
Measure: Mean (Standard Deviation); unit: percentage of time spent < 65 mg/dl
Arm/Group | Basal Insulin, Approved Oral Medications
Number analyzed (Participants) | 26
percentage of time spent < 65 mg/dl | .04 (1.0) [-.6 to 1.4]

3. Secondary Outcome: Change in Percentage of Time Spent at Glycemic Levels >180 mg/dl
Time Frame: Measured at baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage of time spent >180 mg/dl
Arm/Group | Basal Insulin, Approved Oral Medications
Number analyzed (Participants) | 26
percentage of time spent >180 mg/dl | -8.5 (16.9)

4. Secondary Outcome: Change in Basal Insulin Dose From Baseline Values
Time Frame: Assessed at baseline and 6 months
Measure: Mean (Standard Deviation); unit: units of insulin
Arm/Group | Basal Insulin, Approved Oral Medications
Number analyzed (Participants) | 26
units of insulin | 0.3 (16.7)

ADVERSE EVENTS:
Description: 0 serious adverse events were recorded. 3 device related adverse events were recorded.
Arm/Group | Basal Insulin, Approved Oral Medications
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 3/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basal Insulin, Approved Oral Medications (N=30)
Insertion site irritation (Skin and subcutaneous tissue disorders) | 3 (3) — Includes mild irritation at the site of insertion that has been deemed to be device related by the Primary Investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No